CLINICAL TRIAL: NCT04601948
Title: AYActive Study! A Physical Health Activity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucas Carr (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Lucas Carr, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201907702
Record Dates: First submitted 2019-11-18; First posted 2020-10-26 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Cancer
Keywords: Adolescents; Young Adults
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention will include an activity monitor and access to the mHealth physical activity intervention for 6 weeks. The intervention will include regular motivational messages to encourage activity, a social media thread to provide social support, and a series of fun virtual walking races.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will receive a Fitbit activity monitor and access to the mHealth physical activity intervention for 6 weeks. The intervention will include regular motivational messages to encourage activity, a social media thread to provide social support, and a series of fun virtual walking races.
  Interventions: Behavioral: mHealth Activity Intervention

INTERVENTIONS:
Behavioral: mHealth Activity Intervention — Eligible participants will receive a Fitbit activity monitor and access to our mHealth physical activity intervention for 6 weeks. The intervention will include regular motivational messages to encourage activity, a social media thread to provide social support, and a series of fun virtual walking races.

SUMMARY:
The purpose of this pilot study is to explore the feasibility, acceptability, and efficacy of a 6-week mobile health (mHealth) physical activity intervention among adolescent and young adult (AYA) cancer survivors being treated at the University of Iowa Hospitals and Clinics.

DETAILED DESCRIPTION:
The purpose of this pilot study is to explore the feasibility, acceptability, and efficacy of a 6-week mobile health (mHealth) physical activity intervention among adolescent and young adult (AYA) cancer survivors being treated at the University of Iowa Hospitals and Clinics. Eligible participants will receive a Fitbit activity monitor and access to the mHealth physical activity intervention for 6 weeks. The intervention will include regular motivational messages to encourage activity, a social media thread to provide social support, and a series of fun virtual walking races. AYA cancer survivors between 13-39 years are invited to participate and the impact of this intervention will be tested over 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female cancer survivors
* Diagnosed between 13 and 39 years old
* Currently 3-24 months post-treatment (or in maintenance therapy)
* Receiving survivorship care at HCCC/UIHC
* In remission
* Physically able to walk without limitations
* Own a smartphone with a data plan that is also capable of receiving and sending texts
* Able to understand English and provide informed assent/consent

Exclusion Criteria:

* Physically unable to walk without limitations
* Actively receiving cancer treatment
* Does not own a smartphone with a data plan
* Visual or cognitive impairments causing inability to read, complete or sign the consent form and survey
* Participants with diagnosis of thyroid cancer (due to differences in physical, psychological, emotional, and social effects)
* Presence of a psychiatric disorder that is not managed/unstable or suicidal ideation/actuation in preceding 12 months
* Currently meeting physical activity requirements per American Cancer Society guidelines (150 or more minutes per week of moderate to vigorous physical activity)

Ages: 13 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Number of steps taken per day | Dail steps will be measured each day of the intervention for 7 weeks
  Number of steps taken per day on each day of the intervention

SECONDARY OUTCOMES:
PROMIS Fatigue Scale | Change in fatigue over 7 weeks
  8 item scale, lower score is better
PROMISE Pain Scale | Change in pain over 7 weeks
  8 item scale, lower score is better
PROMIS Physical Function Scale | Change in physical function over 7 weeks
  8 item scale, lower score is better
PROMIS Depression Scale | Change in depression over 7 weeks
  8 item scale, lower score is better
PROMIS Anxiety Scale | Change in anxiety over 7 weeks
  8 item scale, lower score is better
Exercise Self-Regulatory Efficacy | Change in exercise self regulatory efficacy over 7 weeks
  20 item scale, higher score is better
Social Support for exercise | Change in social support for exercise over 7 weeks
  13 item scale, higher score is better

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Carr, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No